CLINICAL TRIAL: NCT01480401
Title: The Long Term Effects of Dietary Sodium Restriction on Clinical Outcomes in Patients With Heart Failure
Brief Title: Study of Dietary Intervention Under 100 MMOL in Heart Failure
Acronym: SODIUM-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 82-SH-01
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2022-06-09 (Actual); Status verified 2014-12

CONDITIONS: Heart Failure
Keywords: Patients with stable heart failure
MeSH Terms: conditions — Heart Failure | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low-sodium diet (Experimental): (1500 mg daily)
  Interventions: Other: low-sodium diet (1500 mg daily)
- moderate-sodium diet (No Intervention): sodium (100 mmol or 2300 mg daily; Usual Care)

INTERVENTIONS:
Other: low-sodium diet (1500 mg daily)
  Arms: low-sodium diet

SUMMARY:
This study aims to identify the relationship between a low-sodium diet and neurohormonal and clinical status in stable chronic HF patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be recruited from each research center if they are 18 years or older, with confirmed diagnosis of Heart Failure (including both those with a reduced and preserved systolic function), NYHA II-IV, and willing to sign informed consent.

Exclusion Criteria:

* Subjects will be excluded if they have severe hyponatremia (serum sodium <130 mmol/L)
* Renal failure (a glomerular filtration rate < 30 mL/min)
* Uncontrolled thyroid disorders
* Hepatic failure
* Implantable cardiac device (ICD or CRT) or myocardial revascularization procedures (coronary angioplasty and/or surgical revascularization) in the previous 3 months
* Uncontrolled atrial fibrillation or recurrent ventricular arrhythmias
* Malignancy, or with moderate-severe dementia.
* Patients will be excluded if, in the opinion of the investigator, another condition exists that would preclude dietary compliance or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
composite clinical outcomes | 12 months
  (cardiovascular hospitalizations, emergency department visits due acute decompensated HF, and all-cause mortality) in patients with stable HF

SECONDARY OUTCOMES:
symptoms and quality of life | 12 months
  improves symptoms and quality of life for patients with stable HF
reduces natriuretic peptide levels | 12 months
  reduces natriuretic peptide levels

CONTACTS AND LOCATIONS:
Overall Officials: Justin Ezekowitz, MBBCh MSc, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Colin-Ramirez E, McAlister FA, Zheng Y, Sharma S, Ezekowitz JA. Changes in dietary intake and nutritional status associated with a significant reduction in sodium intake in patients with heart failure. A sub-analysis of the SODIUM-HF pilot study. Clin Nutr ESPEN. 2016 Feb;11:e26-e32. doi: 10.1016/j.clnesp.2015.11.002. Epub 2015 Dec 29. PMID 28531423